CLINICAL TRIAL: NCT03560115
Title: Reliability and Normative Value of Single Heel-rise Test in School-going Children
Brief Title: Normative Value of Single Heel-rise Test in School-going Children Along With Its Inter-session Agreement
Status: Completed | Type: Observational
Sponsor: Asir John Samuel (Other)
Responsible Party: Sponsor-Investigator, Asir John Samuel, Associate Professor, Maharishi Markendeswar University (Deemed to be University)
Organization: Maharishi Markendeswar University (Deemed to be University) (Other)
Other Study IDs: MMDU/IEC/1119; U1111-1214-2525 (Other: Universal Trial Number (UTN))
Record Dates: First submitted 2018-05-18; First posted 2018-06-18 (Actual); Last update posted 2019-03-19 (Actual); Status verified 2019-03

CONDITIONS: Healthy
Keywords: Children; Heel; Reliability

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Single-heel rise test — Single heel-rise test is used to assess the strength of plantar-flexors clinically

SUMMARY:
Background:

Single heel-rise test (SHRT) is a method of assessing the strength and endurance of plantar-flexors manually. Single heel-rise test also known as calf rise test, is a method of assessing the strength of plantar-flexor. The test was first done to determine the integrity of calf muscle. There are few studies which has established the reliability and normative value of heel-rise test in adults. But till date, there is no documented evidence of normative value of heel-rise test in children.

Aim:

The study is focused to derive reliability and normative value of single heel-rise test in children of age group 8-12 years.

Methods:

The study will recruit healthy school-going children of 8-12 years age. Any pathology which can limit or interfere with the test outcome will be excluded. The samples will be collected by stratified sampling technique. Procedure of test will be demonstrated prior to the test. Heel raising and lowering will be performed until child feels fatigue. Test will be performed on both the lower extremities individually.

Data analysis:

Test will be assessed on both the heel individually. Three sessions will be conducted by the same rater on same child for intra-rater and test-retest reliability, and another rater will assess the test on same individual for establishing inter-rater reliability. Normative value of the test will be determined by deriving the mean of test-values for each age group.

DETAILED DESCRIPTION:
1. Introduction:

   Plantar flexors play a crucial role in gait cycle, during foot clearance. It assists in forward propulsion, and is also responsible for maintaining the static and dynamic balances. Single heel-rise test is a physical examination which evaluates the strength of plantar-flexors. This study aims to assess the intra-rater and inter-rater reliability and normative value of single heel-rise test in healthy school-going children of age group 8-12 years.

   1.1.Problem Statement: The documented evidences does not have normative value for single heel-rise test in children. The normative value is provided only for adults. Therefore, there is an absolute need of deriving normative value for this test in children.

   1.2.Purpose of the study: The purpose of this study is to derive the normative value of single-heel rise test along with reliability.

   1.3.Objectives of the study: 1.3.1.To establish inter-rater and intra-rater and test-retest reliability of single heel-rise test 1.3.2.To derive normative value of single heel-rise test
2. Procedure:

The study will be a cross-sectional study. The study protocol has been approved from the Institutional Ethics Committee of Maharishi Markandeshwar (Deemed to be University).

All the anthropometrics of the children will be taken prior to the test which includes height, weight, calf muscle girth and length. The maximum number of heel-rises will be performed by the child in single limb stance until maximal exertion will be recorded. The test will be repeated in standing position on both the sides. For balancing, 2-finger support on wall will be allowed.

Reliability testing: For inter-rater, 2 raters will assess on two different sessions on same day. For intra-rater, same rater will assess the test twice on same day, and after 24 hours for test-retest reliability.

Normative value: The mean of all the test-values for each age group will be normative value for that particular age group.

ELIGIBILITY:
Inclusion Criteria:

* Age group 8-12 years
* Both boys and girls
* Healthy school going children

Exclusion Criteria:

* Un co-operative children
* Children with recent history of injury or surgery in past 6 months
* Any condition that can limit the test outcome (Pain, weakness, etc)

Ages: 8 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: The study will be conducted on healthy children of 8-12 years age group. Any condition that can limit the test measure will be excluded as the test is aimed to achieve normative value.
Sampling Method: Probability Sample
Enrollment: 500 (Actual)
Dates: Start 2018-10-15 (Actual); Primary Completion 2019-01-10 (Actual); Study Completion 2019-03-01 (Actual)

PRIMARY OUTCOMES:
Number of heel raise | Upto two weeks
  Until exhaustion, number of times the heel raise can be achieved by participant

CONTACTS AND LOCATIONS:
Overall Officials: Rajnee Mishra, BPT, (MPT), Principal Investigator — Department of Pediatrics and Neonatal Physiotherapy, MMIPR
Locations (1):
- Maharishi Markandeshwar Institute of physiotherapy and Rehabilitation, Ambāla, Haryana, India

IPD SHARING:
Plan to Share IPD: Undecided
It is yet not decided

REFERENCES:
- [Result] Monteiro DP, Britto RR, Fregonezi GAF, Dias FAL, Silva MGD, Pereira DAG. Reference values for the bilateral heel-rise test. Braz J Phys Ther. 2017 Sep-Oct;21(5):344-349. doi: 10.1016/j.bjpt.2017.06.002. Epub 2017 Jul 3. PMID 28709587
- See also: Reference values for the bilateral heel-rise test — https://doi.org/10.1016/j.bjpt.2017.06.002